CLINICAL TRIAL: NCT03011151
Title: Examining the Role of Protease-activated Receptor 2 Agonists in Gastrointestinal Dysfunction in Pediatric Surgical Critical Illness
Brief Title: Protease Activated Receptor-2 and Gastrointestinal Dysfunction in Critical Illness
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Boston Children's Hospital (Other)
Responsible Party: Principal Investigator, Enid Martinez, Assistant in Critical Care Medicine, Boston Children's Hospital
Other Study IDs: IRB-P00024070
Record Dates: First submitted 2017-01-02; First posted 2017-01-05 (Estimated); Last update posted 2023-03-14 (Actual); Status verified 2023-03

CONDITIONS: Gastroparesis; Gastrointestinal Disorder, Functional; Critical Illness
Keywords: pediatric; critical illness; surgery; gastrointestinal dysfunction; gastric emptying; epithelial barrier; nutrition
MeSH Terms: conditions — Gastroparesis; Gastrointestinal Diseases; Critical Illness

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood, Stool
Oversight: Data Monitoring Committee: No

SUMMARY:
Gastrointestinal (GI) dysfunction affects up to 50% of medical and surgical critically ill children. GI dysfunction, specifically gastric dysmotility and loss of epithelial barrier integrity, is associated with significant morbidity in critical illness. The mechanisms underlying GI dysfunction in critical illness are not well understood. GI dysfunction in surgery and critical illness has been associated with inflammation. There is evidence to suggest the protease-activated receptor 2 (PAR2) is a link between inflammation and GI dysfunction. PAR2 is a G-coupled receptor present throughout the GI tract. PAR2 mediates GI motility and epithelial barrier integrity. PAR2 is activated by PAR2 agonists, specifically GI serine proteases and zonulin, released under conditions of inflammation. In this study the investigators will examine the relationship between inflammation and PAR2 activation by PAR2 agonists and subsequent GI dysfunction in pediatric critically ill surgical patients. The overall hypothesis of this study is that PAR2 activation by PAR2 agonists, GI serine proteases and zonulin, released due to inflammation results in gastric dysmotility and loss of epithelial barrier integrity. In this study, the investigators will examine whether PAR2 agonist expression is increased and correlates with GI dysfunction in critically ill surgical pediatric patients. This proposal fills a knowledge gap in the understanding of mechanisms for GI dysfunction in critical illness, and will be applicable to all surgical and medical critically ill children.

DETAILED DESCRIPTION:
The investigators in this study aim to examine a plausible mechanism by which gastrointestinal dysfunction, gastric dysmotility and loss of epithelial barrier integrity, occur in critical illness. Specifically, the investigators will examine whether an increase in PAR2 agonist levels, zonulin and serine proteases, are associated with gastric dysmotility and loss of epithelial barrier integrity in critical surgical illness in children. The investigators will examine GI function, gastric motility and epithelial barrier integrity, and PAR2 agonist levels, zonulin and serine protease, in participants before surgery and after surgery. Specifically, children undergoing posterior spinal fusion, a known significant inflammatory trigger, and with planned admissions to the intensive care unit will be enrolled. Gastrointestinal function and PAR2 agonist levels will be tested non-invasively in blood and stool.

ELIGIBILITY:
Inclusion Criteria:

* 2 years and older

Exclusion Criteria:

* Liver dysfunction
* Renal dysfunction
* Pre-diagnosed gastroparesis/ delayed gastric emptying
* Pre-diagnosed gastrointestinal malabsorption
* Contraindication to acetaminophen administration

Ages: 2 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Children undergoing posterior spinal fusion and admitted to the pediatric intensive care unit
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2017-08-01 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
PAR2 agonist activity- serum zonulin | Immediately pre-operative versus post-operative day 1
  PAR2 agonist activity will be measured by serum zonulin levels (ng/mL)
PAR2 agonist activity- fecal protease activity | Immediately pre-operative versus post-operative day 1
  PAR2 agonist activity will be measured by fecal serine protease activity (trypsin units/gm protein)

SECONDARY OUTCOMES:
Gastric motility by the acetaminophen absorption test- AUC | Immediately pre-operative versus post-operative day 1
  Pharmacokinetic parameters of acetaminophen will be used to determined gastric motility including the concentration of acetaminophen at 60 minutes (mcg/mL).
Gastric motility by the acetaminophen absorption test- Tmax | Immediately pre-operative versus post-operative day 1
  Pharmacokinetic parameters of acetaminophen will be used to determined gastric motility including the time to maximum concentration of acetaminophen (minutes).
Gastric motility by the acetaminophen absorption test- Cmax | Immediately pre-operative versus post-operative day 1
  Pharmacokinetic parameters of acetaminophen will be used to determined gastric motility including area under the curve at 60 minutes (mcg*min/mL).
Epithelial barrier integrity by serum biomarkers | Immediately pre-operative versus post-operative day 1
  Epithelial barrier integrity by serum biomarkers, specifically serum zonulin (ng/mL) and lipopolysaccharide binding protein levels (ng/mL).

CONTACTS AND LOCATIONS:
Overall Officials: Enid Martinez, MD, Principal Investigator — Boston Children's Hospital
Locations (1):
- Boston Children's Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No